CLINICAL TRIAL: NCT07301944
Title: Adversity as a Factor Associated With the Development of Fibromyalgia in Patients With Rheumatologic Diseases and Healthy Controls
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Principal Investigator, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-5559-25-27-1; IRE-5559-25-27-1 (Registry Identifier: Adversity as a factor associated with the development of fibromyalgia)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with rheumatologic diseases
- Healthy controls

SUMMARY:
Adverse experiences, such as exposure to stressful or traumatic events, have been consistently associated with immune system dysfunction, accelerated inflammatory processes, and an increased risk of developing musculoskeletal symptoms, as well as autoimmune and rheumatologic diseases. The etiopathogenesis of this broad group of conditions is highly complex, involving the interaction of genetic, environmental, hormonal, and immunological factors. Although in many cases no clear external trigger can be identified, scientific evidence has shown that adverse experiences-particularly those occurring during childhood-can induce both acute and chronic stress responses that, over time, disrupt the normal function of the hypothalamic-pituitary-adrenal (HPA) axis. This alteration has been proposed as one of the possible biological explanations for the association described between adversity and the onset of rheumatologic and musculoskeletal disorders.

The primary objective of the present proposal is to evaluate the risk of developing fibromyalgia in relation to the presence of adverse experiences, both in patients already diagnosed with rheumatologic diseases and in healthy individuals. To achieve this objective, a longitudinal follow-up study is proposed in which two cohorts will be systematically evaluated: the first cohort will consist of patients with a confirmed diagnosis of rheumatologic conditions, while the second cohort will consist of healthy individuals, carefully matched to the patient group by age and sex in order to minimize potential confounding factors.

The study will begin with a defined selection period, during which eligibility will be verified according to rigorous inclusion and exclusion criteria. Only those individuals who meet all requirements will be enrolled. After enrollment, comprehensive sociodemographic and clinical data will be collected. Standardized and validated questionnaires will then be administered to explore participants' exposure to adverse experiences, considering both childhood and adulthood events. Additionally, these instruments will be used to assess factors closely linked to overall health outcomes, including quality of life, physical health, and mental health.

Data collection will be performed at multiple time points to capture both baseline and longitudinal information. Specifically, measurements will be obtained at baseline (upon enrollment) and during follow-up assessments at 3, 6, and 12 months. This approach will make it possible to evaluate not only cross-sectional associations but also temporal relationships and dynamic changes over time, thereby providing a more robust understanding of the impact of adverse experiences on the potential development of fibromyalgia.

By integrating clinical and psychosocial data across different time points, the study seeks to clarify the multifactorial mechanisms through which adverse experiences may influence the risk of fibromyalgia among individuals with rheumatologic conditions as well as among healthy participants. Ultimately, the findings may contribute to advancing knowledge about disease risk and progression, with the potential to inform preventive strategies and guide future therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

* Patient who is a beneficiary of institutional care.
* Confirmed diagnosis of rheumatological disease according to the treating physician's criteria.
* Onset of the rheumatological disease in adulthood (>18 years).
* Must have signed the informed consent form to participate in the research study.

Exclusion Criteria Cohort 1:

* Concomitant diagnosis of severe disease that compromises the person's short-to-medium-term survival.
* Diagnosis of fibromyalgia self-reported or confirmed during the selection process.
* Lack of availability for follow-up.

Inclusion Criteria Cohort 2:

Exclusion Criteria Cohort 2:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Patients who are beneficiaries of institutional care, Age $\geq 18$ years, with a diagnosis of a rheumatological disease, who will be followed for 12 months. Questionnaires will be answered on paper or through a digital platform, according to the participant's preference. Cohort 2: Healthy individuals matched for age and sex with patients diagnosed with a rheumatological disease, who will be followed for 12 months. Questionnaires will be answered on paper or through a digital platform, according to the participant's preference.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
Newly Diagnosed Fibromyalgia | From enrollment to the end of the study at 12 months.
  A diagnosis of fibromyalgia will be established for all participants who, over the 12 months of the study, obtain a Widespread Pain Index (WPI) score ≥7 plus a Symptom Severity (SS) Scale score ≥5, OR a WPI score between 3 and 6 plus an SS Scale score ≥9.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Medical Sciences and Nutrition, Salvador Zubiran, Tlalpan, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided